CLINICAL TRIAL: NCT00230178
Title: Evaluation of Single Agent Rasburicase for 5 Days Versus Sequential Treatment With Rasburicase From Day 1 Through 3 Followed by Oral Allopurinol From Day 3 Through 5 (Overlap on Day 3) Versus Single Agent Oral Allopurinol for 5 Days in the Management of Plasma Uric Acid in Adult Patients With Leukemia, Lymphoma, and Solid Tumor Malignancies at Risk for Hyperuricemia and Tumor Lysis Syndrome
Brief Title: Rasburicase Versus Allopurinol in Tumor Patients at Risk for Hyperuricemia and Tumor Lysis Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: International Clinical Development, Clinical Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EFC4978
Record Dates: First submitted 2005-09-28; First posted 2005-09-30 (Estimated); Results first posted 2009-12-31 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2010-01

CONDITIONS: Tumor Lysis Syndrome; Cancer; Hyperuricemia
Keywords: Hyperuricemia; Tumor lysis syndrome; Leukemia; Lymphoma; Myelodysplastic Syndromes; Solid tumor cancers; Solid Tumor cancers with hyperuricemia Hyperuricemia (cancer patients only); Tumor lysis syndrome (cancer patients only)
MeSH Terms: conditions — Tumor Lysis Syndrome; Neoplasms; Hyperuricemia; Leukemia; Lymphoma; Myelodysplastic Syndromes | interventions — rasburicase; Urate Oxidase; Allopurinol

ARMS (3):
- Arm A (Experimental): Rasburicase alone given as a single agent for 5 days
  Interventions: Drug: Rasburicase (SR29142)
- Arm B (Experimental): Rasburicase alone given as a single agent from Day 1 through Day 3, followed by oral allopurinol given from Day 3 through Day 5 (Day 3 is an overlap)
  Interventions: Drug: Rasburicase (SR29142); Drug: Allopurinol
- Arm C (Active Comparator): Oral allopurinol alone given as a single agent for 5 days
  Interventions: Drug: Allopurinol

INTERVENTIONS:
Drug: Rasburicase (SR29142) — 30-min IV infusion
  Arms: Arm A; Arm B
Drug: Allopurinol — Oral administration
  Arms: Arm B; Arm C

SUMMARY:
This is a randomized, multi-center, open-label, parallel group study with three arms:

* Rasburicase alone
* Rasburicase followed by Allopurinol
* Allopurinol alone

The primary objective is to compare the adequacy of control of plasma uric acid concentration and the safety profile among the three arms.

DETAILED DESCRIPTION:
After signing the informed consent and having met the inclusion criteria, patients will be randomized to 1 of the 3 arms and treated for a total duration of 5 days. Patients in all arms will receive chemotherapy beginning 4-24 hours after the first dose of rasburicase or allopurinol.

ELIGIBILITY:
Inclusion Criteria:

1. Meets high risk or at potential risk for tumor lysis syndrome (TLS):

   A patient is at high risk for TLS if he/she presents with:
   * Hyperuricemia of malignancy (plasma uric acid > 7.5 mg/dL);
   * A diagnosis of very aggressive lymphoma/leukemia based on the Revised European-American Lymphoma (REAL) classification of lymphoma/leukemia;
   * Acute myeloid leukemia (AML);
   * Chronic myeloid leukemia (CML) in blast crisis; or
   * High grade myelodysplastic syndrome (refractory anemia with excess blast, chronic myelomonocytic leukemia, and refractory anemia with excess blast in transformation) only if they have > 10% bone marrow blast involvement and are given aggressive treatment similar to AML.

   A patient is at potential risk for TLS if he/she presents with:
   * A diagnosis of aggressive lymphoma/leukemia based on the REAL classification of lymphoma/leukemia plus 1 or more of the following criteria:

     * Lactate dehydrogenase (LDH) >= 2 x upper limit of normal (ULN) (IU/L)
     * Stage III-IV disease
     * Stage I-II disease with at least 1 lymph node/tumor > 5 cm in diameter

   In addition to the above-mentioned eligibility criteria, the patients should have the following criteria:
2. Eastern Cooperative Oncology Group (ECOG) performance status 0-3
3. Age >= 18 years
4. Life expectancy > 3 months
5. Negative pregnancy test (females of child bearing potential) and use of effective contraceptive method (for both males and females). A pregnancy test may be performed on serum or urine human chorionic gonadotropin (HCG).
6. Signed written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2004-04; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: International Clinical Development, Study Director — Sanofi
Locations (15):
- United States (15):
  - Alta Bates Comprehensive Cancer Center, Berkeley, California
  - UCLA Medical Center, Los Angeles, California
  - Rocky Mountain Cancer Center, Denver, Colorado
  - University of Florida Health Science Center at Jacksonville, Jacksonville, Florida
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - New York Methodist Hospital, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - University of Rochester Medical Center, Rochester, New York
  - New York Medical College, Valhalla, New York
  - Duke University Medical Center, Durham, North Carolina
  - Oregon Health and Sciences University, Portland, Oregon
  - University of Pennsylvania Health Systems, Philadelphia, Pennsylvania
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Mary Babb Randolph Cancer Center, Morgantown, West Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Rasburicase: Rasburicase (0.20 mg/kg/day) given as a single agent for 5 days
- Rasburicase + Allopurinol: Rasburicase (0.20 mg/kg/day) given alone as a single agent from Day 1 through Day 3, followed by oral allopurinol (300 mg/day) given from Day 3 through Day 5 (Day 3 is an overlap)
- Allopurinol: Allopurinol (300 mg/day) given alone as a single agent for 5 days
Period: Overall Study
Arm/Group | Rasburicase | Rasburicase + Allopurinol | Allopurinol
Started | 94 (Intent-to-treat (ITT)population: randomized patients) | 93 | 93
Treated | 92 (Modified ITT population: ITT patients with at least 1 dose of study drug) | 92 | 91
Completed | 90 | 86 | 86
Not Completed | 4 | 7 | 7
Not completed — Adverse Event | 1 | 5 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Various other reasons | 3 | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rasburicase | Rasburicase + Allopurinol | Allopurinol | Total
Number analyzed (Participants) | 94 | 93 | 93 | 280
Age, Customized [Number; unit: participants]
  <65 years | 63 | 65 | 69 | 197.0
  >=65 years | 31 | 28 | 24 | 83.0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 42 | 29 | 106.0
  Male | 59 | 51 | 64 | 174.0

OUTCOME MEASURES:

1. Primary Outcome: Plasma Uric Acid Responder
Description: Number of patients responding to treatment defined as plasma uric acid levels at Day 3 through Day 7 <7.5 mg/dl.
Time Frame: Day 3 through Day 7
Measure: Number; unit: Participants
Arm/Group | Rasburicase | Rasburicase + Allopurinol | Allopurinol
Number analyzed (Participants) | 92 | 92 | 91
Participants
  Responder | 80 | 72 | 60
  Non-Responder | 12 | 20 | 31
Statistical Analysis 1: Comparison: Rasburicase vs Allopurinol; Test type: Superiority or Other; p = 0.0009, Wilson's method; Difference in response rate % = 21, 95% CI [8.6 to 32.7]
Statistical Analysis 2: Comparison: Rasburicase + Allopurinol vs Allopurinol; Test type: Superiority or Other; p = 0.0632, Wilson's method; Difference in response rate % = 12.3, 95% CI [-0.9 to 25.0]

2. Secondary Outcome: Plasma Uric Acid
Description: Area under the curve concentration versus time curve extrapolated to infinity (AUC) of plasma uric acid values
Time Frame: Day 1 to Day 7
Population: The analysis was performed on the modified ITT-population with an evaluation of plasma uric acid AUC.
Measure: Mean (Standard Deviation); unit: mg*h/dL
Arm/Group | Rasburicase | Rasburicase + Allopurinol | Allopurinol
Number analyzed (Participants) | 80 | 77 | 72
mg*h/dL | 77.25 (57.17) | 108.05 (70.49) | 646.22 (285.29)
Statistical Analysis 1: Comparison: Rasburicase vs Allopurinol; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 2: Comparison: Rasburicase + Allopurinol vs Allopurinol; Test type: Superiority or Other; p < 0.0001, ANOVA

3. Secondary Outcome: Time to Uric Acid Control
Description: Time from the first dose of study drug to the time at which plasma uric acid concentrations were determined <=7.5 mg/dl, measured -4, 4, 24, 48, 72, 96, 120, and 144 hours after infusion.
Time Frame: Day 1 to Day 7
Population: The analysis was performed on a subgroup of patients from the mITT-population with hyperuricemia immediately prior to the first dose of study drug.
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Rasburicase | Rasburicase + Allopurinol | Allopurinol
Number analyzed (Participants) | 18 | 12 | 16
Hours | 4.1 [4.0 to 4.5] | 4.1 [3.9 to 4.5] | 27.0 [4.0 to 49.0]

ADVERSE EVENTS:
Time Frame: Time from the first study drug intake until a maximum follow-up of 30 days after the last dose of antihyperuricemic treatment.
Description: Reported events are treatment emergent adverse events within the time frame mentioned above.
Arm/Group | Rasburicase | Rasburicase + Allopurinol | Allopurinol
Serious Adverse Events (participants affected / at risk) | 36/92 | 32/92 | 29/91
Other Adverse Events (participants affected / at risk) | 91/92 | 92/92 | 90/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rasburicase (N=92) | Rasburicase + Allopurinol (N=92) | Allopurinol (N=91)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 3 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Multi-organ failure (General disorders) | 2 | 2 | 2
Pyrexia (General disorders) | 2 | 1 | 0
Adverse drug reaction (General disorders) | 1 | 0 | 0
Disease progression (General disorders) | 0 | 1 | 1
Death (General disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0
Neutropenic infection (Infections and infestations) | 5 | 4 | 8
Neutropenic sepsis (Infections and infestations) | 5 | 1 | 3
Sepsis (Infections and infestations) | 1 | 1 | 1
Infection (Infections and infestations) | 1 | 0 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0
Systemic mycosis (Infections and infestations) | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 1
Abdominal abscess (Infections and infestations) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0
Catheter site infection (Infections and infestations) | 0 | 1 | 0
Muscle abscess (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Lobar pneumonia (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1
Sinusitis fungal (Infections and infestations) | 0 | 0 | 1
Drug toxicity (Injury, poisoning and procedural complications) | 1 | 0 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Renal injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Liver function test abnormal (Investigations) | 0 | 1 | 1
Blood pressure increased (Investigations) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Tumor lysis syndrom (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 3
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Neurotoxicity (Nervous system disorders) | 1 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 0
Reversible posterior leukoencephalopathy syndrom (Nervous system disorders) | 1 | 0 | 0
Haemorrhage intracanial (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 1
Neurological symptom (Nervous system disorders) | 0 | 0 | 1
Agitation (Psychiatric disorders) | 1 | 0 | 0
Completed suicide (Psychiatric disorders) | 0 | 0 | 1
Mania (Psychiatric disorders) | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 1 | 1
Renal failure (Renal and urinary disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rasburicase (N=92) | Rasburicase + Allopurinol (N=92) | Allopurinol (N=91)
Thrombocytopenia (Blood and lymphatic system disorders) | 51 | 49 | 48
Neutropenia (Blood and lymphatic system disorders) | 49 | 44 | 45
Anaemia (Blood and lymphatic system disorders) | 31 | 31 | 43
Febrile neutropenia (Blood and lymphatic system disorders) | 19 | 22 | 21
Leukopenia (Blood and lymphatic system disorders) | 15 | 12 | 11
Lymphopenia (Blood and lymphatic system disorders) | 1 | 5 | 1
Tachycardia (Cardiac disorders) | 20 | 23 | 22
Atrial fibrillation (Cardiac disorders) | 6 | 3 | 3
Angina pectoris (Cardiac disorders) | 5 | 4 | 0
Bradycardia (Cardiac disorders) | 1 | 6 | 4
Ear and labyrinth disorder (Ear and labyrinth disorders) | 1 | 7 | 5
Dry eye (Eye disorders) | 0 | 5 | 0
Nausea (Gastrointestinal disorders) | 53 | 56 | 50
Diarrhoea (Gastrointestinal disorders) | 52 | 52 | 51
Vomiting (Gastrointestinal disorders) | 35 | 34 | 28
Constipation (Gastrointestinal disorders) | 25 | 25 | 31
Abdominal pain (Gastrointestinal disorders) | 18 | 31 | 22
Abdominal pain upper (Gastrointestinal disorders) | 10 | 6 | 16
Dyspepsia (Gastrointestinal disorders) | 9 | 7 | 12
Abdominal distension (Gastrointestinal disorders) | 8 | 8 | 12
Haemorrhoids (Gastrointestinal disorders) | 8 | 4 | 3
Flatulence (Gastrointestinal disorders) | 6 | 8 | 7
Proctalgia (Gastrointestinal disorders) | 4 | 5 | 5
Oral pain (Gastrointestinal disorders) | 4 | 4 | 8
Stomatitis (Gastrointestinal disorders) | 3 | 6 | 7
Dysphagia (Gastrointestinal disorders) | 3 | 6 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 3 | 3 | 5
Abdominal discomfort (Gastrointestinal disorders) | 2 | 5 | 7
Dry mouth (Gastrointestinal disorders) | 2 | 5 | 7
Oedema peripheral (General disorders) | 46 | 40 | 39
Pyrexia (General disorders) | 44 | 56 | 51
Chills (General disorders) | 26 | 33 | 33
Mucosal inflammation (General disorders) | 23 | 25 | 24
Fatigue (General disorders) | 19 | 28 | 34
Asthenia (General disorders) | 12 | 12 | 19
Catheter site pain (General disorders) | 9 | 4 | 8
Pain (General disorders) | 8 | 10 | 7
Oedema (General disorders) | 6 | 2 | 6
Catheter site related reaction (General disorders) | 5 | 2 | 4
Catheter site erythema (General disorders) | 5 | 1 | 8
Catheter site haemorrhage (General disorders) | 4 | 1 | 9
Malaise (General disorders) | 3 | 2 | 5
Hyperbilirubinaemia (Hepatobiliary disorders) | 14 | 13 | 7
Sepsis (Infections and infestations) | 10 | 6 | 3
Bacteraemia (Infections and infestations) | 9 | 7 | 16
Pneumonia (Infections and infestations) | 9 | 2 | 7
Cellulitis (Infections and infestations) | 6 | 0 | 4
Oral candidiasis (Infections and infestations) | 5 | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 6 | 7 | 5
Procedural pain (Injury, poisoning and procedural complications) | 5 | 5 | 2
Transfusion reaction (Injury, poisoning and procedural complications) | 4 | 7 | 8
Aspartate aminotransferase increased (Investigations) | 15 | 22 | 20
Blood bilirubin increased (Investigations) | 14 | 11 | 13
Alanine aminotransferase increased (Investigations) | 10 | 25 | 16
Blood creatinine increased (Investigations) | 7 | 8 | 9
Blood alkaline phophatase increased (Investigations) | 6 | 5 | 4
Blood pressure increased (Investigations) | 4 | 5 | 1
Platelet count decreased (Investigations) | 4 | 5 | 6
Blood lactate dehydrogenase decreased (Investigations) | 2 | 7 | 3
Weight decreased (Investigations) | 2 | 6 | 5
Haemoglobin decreased (Investigations) | 2 | 5 | 6
Blood alkaline phosphatase decreased (Investigations) | 1 | 5 | 3
White blood cell count decreased (Investigations) | 1 | 5 | 3
Blood phosphorus increased (Investigations) | 1 | 2 | 7
Hypokalaemia (Metabolism and nutrition disorders) | 35 | 32 | 36
Hypocalcaemia (Metabolism and nutrition disorders) | 31 | 41 | 44
Hyperglycaemia (Metabolism and nutrition disorders) | 27 | 34 | 35
Hypoalbuminaemia (Metabolism and nutrition disorders) | 25 | 24 | 27
Hyponatraemia (Metabolism and nutrition disorders) | 25 | 21 | 23
Anorexia (Metabolism and nutrition disorders) | 20 | 23 | 25
Hypophosphataemia (Metabolism and nutrition disorders) | 16 | 21 | 15
Hypomagnesaemia (Metabolism and nutrition disorders) | 14 | 15 | 14
Fluid overload (Metabolism and nutrition disorders) | 11 | 6 | 3
Hyperphosphataemia (Metabolism and nutrition disorders) | 9 | 14 | 8
Hyperkalaemia (Metabolism and nutrition disorders) | 7 | 4 | 4
Decreased appetite (Metabolism and nutrition disorders) | 5 | 4 | 6
Hypernatraemia (Metabolism and nutrition disorders) | 5 | 3 | 3
Hyperphosphatasaemia (Metabolism and nutrition disorders) | 2 | 7 | 6
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 6 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 12 | 15
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 11 | 9
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 8 | 7 | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 12 | 18
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 8 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 7 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 5
Headache (Nervous system disorders) | 25 | 31 | 33
Dizziness (Nervous system disorders) | 14 | 17 | 19
Lethargy (Nervous system disorders) | 8 | 6 | 3
Dysgeusia (Nervous system disorders) | 6 | 6 | 6
Somnolence (Nervous system disorders) | 5 | 2 | 4
Syncope (Nervous system disorders) | 2 | 2 | 6
Paraesthesia (Nervous system disorders) | 2 | 2 | 5
Sinus headache (Nervous system disorders) | 0 | 5 | 1
Anxiety (Psychiatric disorders) | 22 | 16 | 16
Insomnia (Psychiatric disorders) | 17 | 27 | 34
Confusional state (Psychiatric disorders) | 15 | 12 | 11
Depression (Psychiatric disorders) | 12 | 6 | 13
Agitation (Psychiatric disorders) | 8 | 1 | 4
Hallucination (Psychiatric disorders) | 3 | 3 | 6
Haematuria (Renal and urinary disorders) | 11 | 11 | 13
Dysuria (Renal and urinary disorders) | 8 | 3 | 4
Proteinuria (Renal and urinary disorders) | 6 | 7 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 20 | 18 | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 17 | 15 | 18
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 16 | 14 | 20
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 13 | 19 | 9
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 10 | 8 | 8
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 10 | 6 | 8
Wheezing (Respiratory, thoracic and mediastinal disorders) | 9 | 8 | 8
Rales (Respiratory, thoracic and mediastinal disorders) | 7 | 6 | 9
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 5
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 5 | 7 | 3
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 5
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 5
Rash (Skin and subcutaneous tissue disorders) | 26 | 31 | 30
Petechiae (Skin and subcutaneous tissue disorders) | 16 | 13 | 12
Pruritus (Skin and subcutaneous tissue disorders) | 10 | 10 | 9
Alopecia (Skin and subcutaneous tissue disorders) | 8 | 7 | 11
Erythema (Skin and subcutaneous tissue disorders) | 7 | 8 | 8
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 7 | 3 | 9
Ecchymosis (Skin and subcutaneous tissue disorders) | 5 | 6 | 5
Rash generalised (Skin and subcutaneous tissue disorders) | 4 | 4 | 5
Hypotension (Vascular disorders) | 27 | 24 | 23
Hypertension (Vascular disorders) | 11 | 9 | 9
Reproductive system and breast disorders (Reproductive system and breast disorders) | 10 | 6 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.